CLINICAL TRIAL: NCT01921933
Title: The "OPEN" Study Optiflow PatEncy and MaturatioN
Brief Title: The Optiflow Patency and Maturation Study
Acronym: OPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioconnect Systems, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCS_TP1070
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: End-stage Kidney Disease; End-stage Renal Disease
Keywords: End-stage renal disease; ESRD; AVF; Fistulas
MeSH Terms: conditions — Kidney Failure, Chronic; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optiflow (Experimental): The Optiflow device will be implanted in the upper extremity of Adult end-stage renal disease (ESRD) patients requiring creation of an upper extremity autogenous arteriovenous fistula for dialysis access.
  Interventions: Device: Optiflow

INTERVENTIONS:
Device: Optiflow — The Optiflow device will be implanted in the upper extremity of Adult end-stage renal disease (ESRD) patients requiring creation of an upper extremity autogenous arteriovenous fistula for dialysis access.
  Other Names: Optiflow Anastomotic Connector

SUMMARY:
The objective of this study is to assess the performance and safety of the Optiflow Anastomotic Connector (Optiflow) when used to facilitate the creation of autogenous arteriovenous fistula (AVF) anastomoses.

DETAILED DESCRIPTION:
The investigation is designed as a multi-center, prospective, single-arm, clinical study of the Optiflow performance and safety in a maximum of 180 subjects which includes one (1) roll-in subjects per investigator (maximum of 36 roll-in subjects). Subjects will be followed at 14 days post-procedure, 42 days post-procedure, and 90 days post-procedures.

Results will be compared to a pre-established performance goal.

Up to fifteen (15) investigational sites will participate in the investigational study.

The primary performance endpoint is the overall maturation percentage rate at 90 days. Maturation is defined as an access site which achieves a diameter of greater or equal to 4 mm and blood flow greater or equal t0 500 mL/min as measured via duplex ultrasound.

The primary safety endpoint is a composite endpoint of serious adverse events known to be associated with arteriovenous fistula anastomosis surgical procedures through 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (verified with a urine/blood pregnancy test, for women of reproductive age).
* Life expectancy of at least one year, per the investigator's opinion.
* Diagnosed with ESRD or chronic kidney disease requiring dialysis.
* Planned upper extremity autogenous arteriovenous fistula.
* Planned anastomosis is an end of vein to side of artery configuration.
* AVF target artery and vein inner diameters are greater or equal to 3.0 mm and less than or equal to 7.0 mm as determined by pre-operative ultrasound and confirmed intra-operatively.
* Patient is available and willing to return for follow-up visits during the duration of the study.
* Patient is able and willing to follow a daily aspirin and/or other anticoagulation/antiplatelet regimen not including warfarin (see exclusion criteria).
* Patient, or their legal representative, is willing and able to provide informed consent.

Exclusion Criteria:

* Known bleeding diathesis or coagulation disorder.
* Documented or suspected central venous stenosis.
* Uncontrolled hypotension with systolic blood pressures < 100 mg Hg at the time of screening.
* Peripheral white blood cell count < 1.5 K/mm3 or platelet count < 75,000 cells/mm3.
* Body Mass Index (BMI) > 42.
* Transposition of the access vein is anticipated within the 90 day follow-up interval.
* Receiving anticoagulant therapy for non-cardiac indications.
* Evidence or history of an active or suspected infection within one month of screening.
* Scheduled kidney transplant within six months of enrollment.
* History of ≥ 2 AVF and/or synthetic access graft failures.
* History of steal syndrome from a previous hemodialysis vascular access which required intervention or abandonment.
* Current participation in another clinical trial (excluding retrospective studies or studies not requiring a consent form).
* Anticipated surgery requiring general anesthesia during the course of follow-up.
* A history of substance abuse.
* Anticipated to be non-compliant with medical care or study requirements based on investigator judgment.
* Need for immunosuppressive therapy at a dose greater than the equivalent of prednisone 10 mg per day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Fistula Maturation | 90 days
  The primary performance endpoint is the maturation percentage rate at 90 days. Maturation is defined as an access site intended for dialysis needle cannulation which achieves a diameter of greater or equal to 4 mm and blood flow greater or equal to 500 mL/min as measured via duplex ultrasound.
Serious Adverse Events Associated with Arteriovenous Fistula Creation | 90 days
  The primary safety endpoint is a composite endpoint of serious adverse events known to be associated with arteriovenous fistula anastomosis surgical procedures through 90 days. All patients will be followed for safety for the duration of the study.

SECONDARY OUTCOMES:
Technical success | 1 day
  Technical success rate: An access site that demonstrates physical exam patency through hospital discharge.
Assisted Maturation | 90 days
  Assisted maturation rate: An access site which achieves or maintains maturation following intervening manipulations (surgical or endovascular) designed to promote or reestablish maturation.
Unassisted Maturation | 90 days
  Unassisted fistula maturation rate: An access site that achieves and maintains maturation without any surgical or endovascular intervention designed to promote or reestablish Maturation.
Assisted Patency | 90 days
  Assisted patency rate: An access site which is patent after intervening manipulations (surgical or endovascular) intended to promote or reestablish patency.
Unassisted Patency | 90 days
  Unassisted patency rate: An access site that maintains patency without any surgical or endovascular intervention designed to maintain or reestablish blood flow in the access site.
Intervention Rate | 90 days
  Intervention rate: The number of occurrences that a subject's access site is surgically or endovascularly operated on to maintain or reestablish blood flow in the access site.

OTHER OUTCOMES:
Time to first cannulation | Up to 90 days
  Elapsed time to first use of access site.
Ultrasound flow | 90 days
  Flow rate of blood through outflow vein
Time To Access Site Abandonment | Up to 90 days
  Elapsed time to abandonment of the access site.
Access Site Related Adverse Events | 90 days
  The number of access related adverse events per subject
Number of Access Site Related Hospitalizations | 90 days
  The number of access site related hospitalizations per subject.
Catheter Utilization | 90 days
  Total number of days a catheter was used before access site maturation per subject.
Total Adverse Events | 90 days
  Total number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati - Division of Nephrology, Cincinnati, Ohio, United States